CLINICAL TRIAL: NCT02090127
Title: Expanded Access Protocol to Provide Ficlatuzumab to P05538 Patient 0001-000412
Brief Title: Protocol to Allow Continued Access of Ficlatuzumab to P05538 Patient
Status: No longer available | Type: Expanded Access
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AV-299-13-103S
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Mullerian Mixed Tumor of Ovary
MeSH Terms: interventions — ficlatuzumab

INTERVENTIONS:
Drug: ficlatuzumab — humanized anti-hepatocyte growth factor (HGF) monoclonal antibody IV administration at 16.5mg/kg every 2 weeks with a ±2 day window around dosing dates, as long as subject is deriving clinical benefit as determined by the Investigator
  Other Names: AV-299; SCH 900105

SUMMARY:
Protocol to Allow Continued Access of Ficlatuzumab to P05538 Patient

DETAILED DESCRIPTION:
This treatment protocol will serve as a mechanism to continue to provide ficlatuzumab to patient 0001-000412, who was previously enrolled under protocol P05538 and whom the investigator believes is deriving clinical benefit from ficlatuzumab treatment.

ELIGIBILITY:
Inclusion Criteria:

* Per original P05538 protocol

Exclusion Criteria:

* Per original P05538 protocol

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- START, San Antonio, Texas, United States

REFERENCES:
- See also: Continued Access of Ficlatuzumab to P05538 Patient — http://clinicaltrials.gov/show/NCT00725634